CLINICAL TRIAL: NCT01367119
Title: A Randomized Comparison of Ketamine and Methohexital Anesthesia for Electroconvulsive Therapy (ECT) in Depression
Brief Title: Ketamine Anesthesia in Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Keith Rasmussen, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-001430
Record Dates: First submitted 2011-06-01; First posted 2011-06-06 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: Depression; Electroconvulsive therapy; Ketamine; Methohexital
MeSH Terms: conditions — Depression | interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Subjects were dosed with approximately 1.0 mg/kg, using ketamine as anesthetic prior to electroconvulsive therapy (ECT).
  Interventions: Drug: Ketamine
- Methohexital (Active Comparator): Subjects were dosed with approximately 1.0 mg/kg, using methohexital as anesthetic prior to electroconvulsive therapy.
  Interventions: Drug: methohexital

INTERVENTIONS:
Drug: Ketamine — Subjects were dosed with approximately 1.0 mg/kg, using ketamine as anesthetic.
  Other Names: Ketalar; Ketamine Hydrocholoride
  Arms: Ketamine
Drug: methohexital — Subjects were dosed with approximately 1.0 mg/kg, using methohexital as anesthetic.
  Other Names: Brevital Sodium
  Arms: Methohexital

SUMMARY:
Does the use of ketamine as the anesthetic medication in electroconvulsive therapy (ECT) accelerate the antidepressant effect of ECT?

The study hypothesis was that depressed subjects receiving ECT with ketamine as the anesthetic agent would demonstrate a faster rate of improvement, defined as lower depression ratings after the second ECT than depressed patients receiving ECT with the usual anesthetic agent.

DETAILED DESCRIPTION:
There are several drugs available to induce anesthesia for electroconvulsive therapy (ECT), a psychiatric treatment for major depressive illness. The most commonly utilized of these include methohexital, thiopental, etomidate, and propofol. Recently, there has been interest in the use of ketamine in sub-anesthetic doses to treat major depressive illness.

In this randomized, blinded trial, depressed subjects scheduled to be treated with ECT were anesthetized with either ketamine or methohexital at doses of approximately 1.0 mg/kg for each drug. Patients received the same drug for up to six of their ECT treatments. Outcome measures included assessments of depressive severity, cognition, post-anesthesia side effects, and hemodynamics.

Subjects were to be followed with as long as they were receiving inpatient ECT treatments. The number of treatments was determined entirely by their primary psychiatric team, also blind to anesthetic, as per usual care. In other words, this study did not determine when to terminate the ECT course.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of depression, either unipolar or bipolar
* Subjects receiving ECT at the Mayo Clinic

Exclusion criteria:

* Subjects not giving their own consent to ECT
* Subjects with schizophrenia, schizoaffective disorder, or dementia
* Subjects diagnosed with a major neurological disorder such as epilepsy, Parkinson disease, multiple sclerosis, or a neurodegenerative dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Rasmussen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic, Rochester, Minnesota.
Period: Overall Study
Arm/Group | Ketamine | Methohexital
Started | 21 | 17
Completed | 19 | 16
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Methohexital | Total
Number analyzed (Participants) | 21 | 17 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 46.95 (13.17) | 48.65 (7.20) | 47.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Depression Rating Using the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 42 (severe symptoms) for either anxiety or depression.
  The questionnaire was administered to the subjects prior to the first treatment, the morning of the third treatment, the morning of the fifth treatment, and the morning of the seventh treatment. For subjects whose treatment series ws cancelled prior to a scheduled next administration of the rating scale, every effort was made to administer them 2 days after the last treatment.
  Means are reported overall across all treatments; p-values also take into account variability across treatments and within subject.
Time Frame: Baseline and after every second treatment for 7 treatments
Population: Analysis was intent to treat; for the ketamine arm there were 54 observations, for the methohexital arm there were 55 observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 21 | 17
units on a scale | 22.08 (8.11) | 24.45 (7.70)
Statistical Analysis 1: Comparison: Ketamine vs Methohexital; P-values take into account variability across treatments and within subject; Test type: Superiority or Other; p = 0.171, t-test, 2 sided

2. Secondary Outcome: Mean Depression Rating Using the Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 27 (severe symptoms) for depression.
  The questionnaire was administered to the subjects prior to the first treatment, the morning of the third treatment, the morning of the fifth treatment, and the morning of the seventh treatment. For subjects whos treatment series ws cancelled prior to a scheduled next administration of the rating scale, every effort was mde to administer them 2 days after the last treatment.
  Means are reported overall across all treatments; p-values also take into account variability across treatments and within subject.
Time Frame: Baseline and after every second treatment for 7 treatments
Population: Analysis was intent to treat; for the ketamine arm there were 65 observations, for the methohexital arm there were 63 observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 21 | 17
units on a scale | 15.98 (7.54) | 17.57 (6.96)
Statistical Analysis 1: Comparison: Ketamine vs Methohexital; P-values take into account variability across treatments and within subject; Test type: Superiority or Other; p = 0.258, t-test, 2 sided

3. Secondary Outcome: Mean Post Anesthesia Recovery Side Effects
Description: Post anesthesia recovery side effects were assessed at the time of discharge from recovery with five patient self-report items: nausea, headache, myalgia, visual disturbance, and confusion. These were rated by the patients on a four point scale (0, 1, 2, 3) - absent, mild, moderate, severe. This means that for each item a subject could score between 0 (no symptoms) and 3 (severe symptoms). Also, degree of recovery room agitation was rated by the nurse on a similar four point scale.
Time Frame: Time of discharge from recovery after ECT for each treatment, approximately 30 minutes after the end of the seizure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 21 | 17
units on a scale
  Nausea | 0.12 (0.39) | 0.15 (0.42)
  Headache | 0.29 (0.61) | 0.35 (0.67)
  Myalgia | 0.07 (0.30) | 0.15 (0.48)
  Visual Disturbance | 0.08 (0.28) | 0.01 (0.11)
  Confusion | 0.70 (0.95) | 0.30 (0.53)
  Recovery Room Agitation | 0.07 (0.26) | 0.09 (0.36)
Statistical Analysis 1: Comparison: Ketamine vs Methohexital; Comparison between groups for nausea; Test type: Superiority or Other; p = 0.091, t-test, 2 sided
Statistical Analysis 2: Comparison: Ketamine vs Methohexital; Comparison between groups for headache; Test type: Superiority or Other; p = 0.763, t-test, 2 sided
Statistical Analysis 3: Comparison: Ketamine vs Methohexital; Comparison between groups for myalgia; Test type: Superiority or Other; p = 0.356, t-test, 2 sided
Statistical Analysis 4: Comparison: Ketamine vs Methohexital; Comparison between groups for visual disturbance; Test type: Superiority or Other; p = 0.093, t-test, 2 sided
Statistical Analysis 5: Comparison: Ketamine vs Methohexital; Comparison between groups for confusion; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 6: Comparison: Ketamine vs Methohexital; Comparison between groups for recovery room agitation; Test type: Superiority or Other; p = 0.860, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Ketamine | Methohexital
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No